CLINICAL TRIAL: NCT06673173
Title: Patient Satisfaction and Oral Health-Related Quality of Life of Quadrilateral Versus Bilateral Linear Bar Designs for Four Implant Implant-Assisted Complete Mandibular Overdenture Regarding Peri-Implant Crestal Bone Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Wageh Abozaed Elsaed Mansour, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: A0101024RP
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Edentulism
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 quadrilateral bar design (Experimental): Quadrilateral Group: each participant received bar mandibular overdentures on 4 implants with quadrilateral distribution. A plastic ready-made bar was cast in cobalt chrome alloy.
  Interventions: Other: Implant
- group2 : Bilateral linear bar (Experimental): Bilateral linear Group: each participant received bar mandibular overdentures on 4 implant on bilateral configuration
  Interventions: Other: Implant

INTERVENTIONS:
Other: Implant — A long cone paralleling approach with a specially made film holder will be used to assess each patient's vertical marginal bone loss to ensure standardized radiography analysis and avoid any magnification errors. The linear distance between the proximal crestal bone level and the implant shoulder will be measured at the mesial and distal aspects of the implant measured in millimeters (mm). Measurements will performed using image measurement software patient satisfaction comparison between 2 groups

SUMMARY:
For this study, twenty patients were selected, and participants were randomly divided into two groups using random numbers produced in an Excel spreadsheet. Each patient got four implants in the mandibular canine and first molar sites, as well as the bar attachment.

The purpose of this study was to document and report patient satisfaction with mandibular implant overdentures with quadrilateral distribution and linear distribution. The null hypothesis was that patient satisfaction would not be different depending on the distribution type (quadrilateral or linear).

According to the bar design, all patients were classified into two equal groups: quadrilateral bar design (group I) and bilateral linear bar design (group II). Peri-implant marginal bone loss was evaluated immediately (T0) and after 2 years (T2) of overdenture insertion using a digital periapical X-ray.

ELIGIBILITY:
Inclusion Criteria:

* have Angle's class I maxilla-mandibular relation
* sufficient inter-arch space
* a healthy, firm mucosa,
* enough residual alveolar ridges in the mandibular regions to support implants

Exclusion Criteria:

* neuromuscular disorder,
* excessive smoking,
* alcoholism,
* parafunctional habits
* systemic disorders affecting the bones
* history of head and neck radiation therapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
marginal bone loss | Peri-implant marginal bone loss was evaluated immediately (T0) and after 2 years (T2) of overdenture insertion using a digital periapical X-ray.
Patient Satisfaction | Patient satisfaction (primary outcome) was measured by a visual analog scale (VAS). OHRQoL (secondary outcome) was measured by oral health impact profile (OHIP-14). Questions of VAS and OHIP-14 were evaluated after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Abozaed, phd, Principal Investigator — Cairo University
Locations (1):
- Heba Wageh Abozaed, Al Mansurah, Egypt